CLINICAL TRIAL: NCT04242628
Title: Social Experiment on the Impact of Social Networking Sites (SNSs) Use on Older People's Wellbeing
Brief Title: The Ageing in a Networked Society -Social Experiment Study
Acronym: ANS-SE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Fondazione Golgi Cenci (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0946
Record Dates: First submitted 2019-12-16; First posted 2020-01-27 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-04

CONDITIONS: Loneliness; Social Isolation
Keywords: UCLA Version 3 scale; LSNS-6 scale
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: The intervention consists of the attendance to two training courses. T1 study members attended a three week course (two classes per week) on smartphones and SNS use. T2 study members attended 5 interactive 90-min meetings on lifestyle education and brain functioning in older people. A goodbye tea was offered after T2 meetings. Throughout the duration of the intervention, we put C study members on a waiting list; at the end of the intervention, in June 2019, interested group C study members attended the SNSs course (held on June 2019). One year after the first intervention, i.e. in March 2020, we will carry out a follow up assessment on T1 and T2 participants. Note that, due to the constraints imposed by the ethical committee (i.e. we offered members of the C group the possibility to attend the SNS course during the first intervention), the members of the C group are excluded from the follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facebook course (Experimental): T1 study members attended a three week course (two classes per week) on smartphones and SNS use. Specifically, the course covers the following topics: smartphone use; Facebook use; WhatsApp use, privacy rules and fraud risk prevention using Facebook. Throughout the duration of the intervention, a tutor was available every Tuesday and Thursday to assist T1 participants in using SNSs.
  Interventions: Other: Facebook course
- Lifestyle course (Experimental): T2 study members attended 5 interactive 90-min meetings on lifestyle education and brain functioning in older people. These meetings covered the following topics regarding good habits for wellbeing at older age: nutrition, brain ageing, physical activity, leisure activities, resources of the city for older people. A goodbye tea was offered after the meetings.
  Interventions: Other: Lifestyle Course
- Waiting list (No Intervention): Throughout the duration of the intervention, we put C study members on a waiting list; at the end of the intervention, in June 2019, interested group C study members attended the SNSs course (held on June 2019).

INTERVENTIONS:
Other: Facebook course — The intervention consists of the attendance to a course on Facebook and Social Networking Sites use
  Arms: Facebook course
Other: Lifestyle Course — The intervention consists of the attendance to a course on lifestyle education and brain functioning in older people
  Arms: Lifestyle course

SUMMARY:
The Ageing in a Networked Society -Social Experiment study (ANS-SE) is a randomised controlled trial on older people residing in Abbiategrasso, a middle-size city located in the Milan area (Italy) and aims to assess the impact of SNS use on loneliness, that is the primary outcome of this study. The study is constituted of two stages, i.e. the baseline and the follow up. The experiment is structured into two treatment groups and a control group; the interventions are the attendance to a course on SNS use (T1) and lifestyle education and brain functioning (T2). The control group (C) is constituted of a waiting list. The study is part of the project "Aging in a networked society. Older people, social networks and well-being", funded by the Italian Fondazione Cariplo.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the short-term and long-term impact of Facebook use on physical and mental health of older people. The experiment is carried out on 180 participants of the Brain Aging in Abbiategrasso Study (InveCe).The InveCE study is a biannual cohort study of older people born between 1935 and 1939 and living in Abbiategrasso, a town near Milan, in northern Italy (NCT01345110, ClinicalTrials.gov). For more information, see http://www.golgicenci.it/en/studio-invece/.

Participants are selected among those who agreed to take part in the 4th wave of the InveCe.Ab study. Inclusion and exclusion criteria are specified in the Eligibility box below. The study is constituted of two stages, i.e. the baseline and the follow up. The experiment is structured into two treatment groups and a control group; the interventions are the attendance to a course on SNS use (T1) and lifestyle education and brain functioning (T2). The control group (C) is constituted of a waiting list. Participant are assigned to one of these three groups randomly. Before/after the intervention, researchers administered a questionaire to participants to measure levels of loneliness, depression and neuropsychological functioning (see the box "Outcome Measure" for the description of the scales and measures used), together with a medical examination. The same assessment will be performed after one year. Data collected will be analyzed using statistical techniques in order to evaluate the impact of Facebook use on well-being.

The study is part of the project "Aging in a networked society. Older people, social networks and well-being", funded by the Italian Fondazione Cariplo.

ELIGIBILITY:
Inclusion Criteria:

* Participants to the third follow-up of the Brain Ageing in Abbiategrasso Study (InveCe.Ab study)
* Good mental health
* No physical limitations
* Good cognitive health
* No experience in using Social Networks SItes (SNSs)

Exclusion Criteria:

* GDS (Geriatric Depression Score) score equal to or greater than 10 (no major depression)
* Hands functional limitations
* Visual or hearing impairment
* Dementia or Mild Cognitive Impairment (MCI),
* Mini-Mental State Examination (MMSE) lower than 24
* Used SNS at least one time in life

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Subjective feeling of loneliness | Change from basline score at UCLA Loneliness Scale at 2 months
  Indicates self feeling of loneliness. Measured with UCLA Loneliness Scale Minimum score: 20; Maximum score: 80 Highest scores indicate greater loneliness (Russell, 1996).
Stroop Test (inhibitory control and cognitive flexibility) | Change from basline score at test at 2 months
  Executive Cognitive Functions measured through the Stroop Test Interference score for time and errors (higher scores worse performance) Score range: n.a. (Cafarra et al., 2002)
Executive Cognitive functions: processing speed in Symbol Search | Change from basline score at test at 2 months
  Executive Cognitive Functions measured through the Digit Symbol test from the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV).
  Symbol Search, score range 0-60 Higher scores better performances (Orsini & Pezzuti, 2013)
Executive Cognitive functions: processing speed in Coding | Change from basline score at test at 2 months
  Executive Cognitive Functions measured through the Digit Symbol test from the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV).
  Coding: score range 0-135 Higher scores better performances (Orsini & Pezzuti, 2013)
Executive Cognitive functions: working memory | Change from basline score at test at 2 months
  Executive Cognitive Functions measured through the Digit Symbol test from the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV).
  Digit Span: score range 0-48 Higher scores better performances (Orsini & Pezzuti, 2013)
Executive Cognitive Functions - Trail Making Test (TMT) | Change from basline score at test at 2 months
  Executive Cognitive Functions measured through the Trail Making Test (TMT) (Giovagnoli et al., 1996)
Cumulative Illness Rating Scale | Change from basline score at scale at 2 months
  Clinical tool to measure objective older people illness status Scores range between 14 to 70 with a higher score indicating worse health satus (Parmelee et al. 1995)
Blood Pressure | Change from basline score for blood pressure at 2 months
  High blood pressure, measured in mmHg,can be an indicator of stress or other health problems
6 items Lubben Social Network Scale | Change from basline score at Lubben Social Network scale at 2 months
  This scale is a self-report measure of social engagement including family and friends. The score ranges between 0 and 30, with a higher score indicating more social engagement. (Lubben et al. 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Sala, PhD, Principal Investigator — Università degli Studi di Milano-Bicocca
Locations (1):
- Fondazione Golgi Cenci, Abbiategrasso, Milano, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request by email to Fondazione Golgi Cenci. Applicants will receive a form to fill with all the information about the research design and purpose. The application will be evaluated by a comittee chaired by Prof. Emanuela Sala. The final decision will be communicated within two weeks.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from November 2020 without a deadline
Access Criteria: Data available upon written request by email to Fondazione Golgi Cenci (check the following URL)
URL: http://www.golgicenci.it/contatti/

REFERENCES:
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Giovagnoli AR, Del Pesce M, Mascheroni S, Simoncelli M, Laiacona M, Capitani E. Trail making test: normative values from 287 normal adult controls. Ital J Neurol Sci. 1996 Aug;17(4):305-9. doi: 10.1007/BF01997792. PMID 8915764
- [Background] Caffarra P., Vezzadini G., Dieci F., Zonato A., Venneri A., Una versione abbreviata del test di stroop: dati normativi nella popolazione italiana. Nuova Rivista di Neurologia 2002, 12 (14): 111-115.
- [Background] Parmelee PA, Thuras PD, Katz IR, Lawton MP. Validation of the Cumulative Illness Rating Scale in a geriatric residential population. J Am Geriatr Soc. 1995 Feb;43(2):130-7. doi: 10.1111/j.1532-5415.1995.tb06377.x. PMID 7836636
- [Background] Orsini A., Pezzuti L.(2013). WAIS-IV. Contributo alla taratura italiana.Giunti OS. Firenze.
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Derived] Rolandi E, Vaccaro R, Abbondanza S, Casanova G, Pettinato L, Colombo M, Guaita A. Loneliness and Social Engagement in Older Adults Based in Lombardy during the COVID-19 Lockdown: The Long-Term Effects of a Course on Social Networking Sites Use. Int J Environ Res Public Health. 2020 Oct 28;17(21):7912. doi: 10.3390/ijerph17217912. PMID 33126634
- See also: Fondazione Golgi Cenci — http://www.golgicenci.it/
- See also: Fondazione Cariplo — http://www.fondazionecariplo.it/it/index.html
- See also: Ethical Committee (Università Bicocca) — https://www.unimib.it/ricerca/comitato-etico
- See also: PI's University page — https://www.unimib.it/emanuela-maria-sala
- See also: Brain ageing in Abbiategrasso study — http://www.golgicenci.it/studio-invece/